CLINICAL TRIAL: NCT06825676
Title: Guideline-diRected MAnagement for Chronic Kidney Disease: EValuation of an Education Progamme in a National Cluster Randomized Controlled Trial (GRAVER)
Brief Title: Guideline-diRected MAnagement for Chronic Kidney Disease: EValuation of an Education Progamme in a National Cluster Randomized Controlled Trial
Acronym: GRAVER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Principal Investigator, Jiyan Chen, professor, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Guangdong Provincial People's
Record Dates: First submitted 2025-02-09; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Renal Insufficiency, Chronic; Cardiovascular Diseases (CVD)
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Masking Description: Research Statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care Group (No Intervention): Participants in the control group will receive the usual care protocol. Healthcare personnel at the control center only receive routine community training without additional medical education interventions. These healthcare personnel provide routine diagnosis and treatment to patients as well as subsequent follow-up.
- CKD Patient Management Based on Guidelines (Active Comparator): The intervention group will implement comprehensive management for CKD patients based on guidelines, including lifestyle education, pharmacological treatment, risk factor management, risk assessment, referral management, and the completion of the CKD patient management checklist.
  Interventions: Behavioral: CKD Patient Management Based on Guidelines

INTERVENTIONS:
Behavioral: CKD Patient Management Based on Guidelines — 1. Lifestyle Education: smoking cessation, physical activity, healthy eating, and weight management.
  2. Pharmacological Treatment: Implement targeted and guideline-based pharmacological treatment plans for patients with different comorbidities, such as the use of RAAS inhibitors (RASi), SGLT2 inhibitors, statins, and other medications.
  3. Risk Factor Management: Effectively manage risk factors such as hypertension, diabetes, and dyslipidemia, and regularly reassess these factors.
  4. Risk Assessment: Perform risk assessments for CKD patients based on eGFR and UACR, and implement graded management according to the results.
  4、Referral Management: Refer patients with eGFR < 30 ml/min/1.73m² or severe proteinuria.
  5、CKD Patient Management Checklist: Community doctors should complete the CKD patient management checklist in a standardized manner, including records of risk factors, dynamic kidney function, and follow-up plans.
  Arms: CKD Patient Management Based on Guidelines

SUMMARY:
Study Objective:

To evaluate the impact of guideline-based CKD comprehensive management medical re-education for community healthcare providers on improving cardio-renal outcomes in CKD patients.

Study Design:

A nationwide, multicenter, prospective, cluster-randomized controlled trial.

Inclusion and Exclusion Criteria:

Inclusion Criteria: Chronic kidney disease (CKD) patients meeting the following criteria:

eGFR <60 mL/min/1.73 m² or UACR >30 mg/g on two separate occasions at least 3 months apart.

Exclusion Criteria:

Age <18 years. End-stage renal disease (ESRD) with eGFR <15 mL/min/1.73 m², or patients already on regular dialysis or having received a kidney transplant.

Pregnant or breastfeeding women. Patients participating in any other clinical trials. Patients who exhibit characteristics at the screening stage that suggest they are unable to complete the study.

Intervention:

Control Group: Routine community training and management. Intervention Group: Training for community healthcare providers on guideline-based CKD management, including lifestyle management, risk assessment and referral recommendations, risk factor control, pharmacological treatment, and the application of a CKD management checklist incorporating these components.

Efficacy Evaluation Indicators:

Primary Outcome:

A renal composite endpoint, defined as at least a 25% decline in eGFR, progression to ESRD (dialysis, kidney transplantation, or sustained eGFR <15 mL/min/1.73 m²), or death due to renal or cardiovascular causes.

Secondary Outcomes:

Cardiovascular composite endpoint: cardiovascular death, non-fatal stroke, non-fatal myocardial infarction, and hospitalization for heart failure.

Delayed CKD progression, defined as a reduction in the annual eGFR decline rate by 0.5-1 mL/min/1.73 m² or a 30% reduction in UACR per year.

Proportion of patients receiving guideline-recommended pharmacological treatment.

Safety Evaluation Indicators:

Acute deterioration of renal function (serum creatinine increase >30% within 4 weeks).

New-onset hyperkalemia. Symptomatic hypotension. Recurrent hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

Patients with chronic kidney disease (CKD) (defined as eGFR <60 ml/min/1.73 m² or UACR >30 mg/g on two occasions at least 3 months apart).

Exclusion Criteria:

1. Age <18 years
2. Patients with end-stage renal disease (eGFR <15 ml/min/1.73 m²) or those already receiving regular dialysis or kidney transplantation
3. Pregnant or breastfeeding women
4. Patients currently participating in any other clinical trial
5. Patients who exhibit characteristics during the screening phase that indicate an inability to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
The renal composite endpoint | 2 years
  a decline in eGFR of at least 25%, end - stage renal disease (including dialysis, kidney transplantation, or eGFR sustained at <15 ml/min/1.73 m²), or death from renal/cardiovascular causes

SECONDARY OUTCOMES:
The cardiovascular composite endpoint | 2 years
  cardiovascular death, non-fatal stroke, non-fatal myocardial infarction, and hospitalization for heart failure
The delay in renal function progression in participants | 2 years
  a decline in eGFR slope of 0.5-1.0 mL/min/1.73 m² per year or a reduction in uACR of 30% per year
The proportion of patients receiving guideline - based pharmacological treatment | 2 years
  The proportion of patients receiving guideline - based pharmacological treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China